CLINICAL TRIAL: NCT05779072
Title: MiSight Lens Wear Cessation Study
Brief Title: Dual Focus Soft Contact Lens Wear Cessation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MIST-402
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-03

CONDITIONS: Myopia
Keywords: Myopia Control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dual Focus for 3 years (Other): Group of subjects who completed dual focus soft contact lens wear treatment for 3 years
  Interventions: Device: Single Vision Soft Contact Lens
- Dual Focus for 6 years (Other): Group of subjects who completed dual focus soft contact lens wear treatment for 6 years
  Interventions: Device: Single Vision Soft Contact Lens

INTERVENTIONS:
Device: Single Vision Soft Contact Lens — Subjects refit to Single Vision Soft Contact Lens for 1 year

SUMMARY:
The purpose of this study is to investigate the effect of ceasing treatment with dual focus soft contact lenses.

DETAILED DESCRIPTION:
This is a bilateral, open label, dispensing study with subjects who have completed dual focus soft contact lens wear treatment for either 3 or 6 years and who are refit to Proclear 1-day lens for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed the MIST-401 Parts 1 and 2
* Visual acuity (VA) with CLs better than +0.25 log MAR (>6/12 or >20/40) in both eyes
* No ocular pathology or other contraindication to contact lens wear
* Where applicable (dependent on local requirements), have:

  1. read the Informed Assent
  2. been given an explanation of the Informed Assent,
  3. indicated an understanding of the Informed Assent and
  4. signed the Informed Assent Form. Or
  5. read the Informed Consent,
  6. been given an explanation of the Informed Consent,
  7. indicated an understanding of the Informed Consent and
  8. signed the Informed Consent Form.
* Where applicable (dependent on local requirements), have their parent or legal guardian:

  1. read the Informed Consent,
  2. been given an explanation of the Informed Consent,
  3. indicated an understanding of the Informed Consent and
  4. signed the Informed Consent Form.
* Along with their parent or guardian (if applicable), be capable of comprehending the nature of the study, and be willing and able to adhere to the instructions set forth in this protocol.
* Along with their parent or guardian (if applicable), agree to maintain the visit schedule and be able to keep all appointments as specified in the study protocol for the duration of the study.
* Agree to wear the assigned contact lenses for a minimum of 10 hours per day, at least 6 days per week, for the duration of the study and to inform the study investigator if this schedule is interrupted. (Wearing time may be modified by the study staff for health reasons.)
* Be in good general health, based on his/her and parent's/guardian's (if applicable) knowledge.
* Have best-corrected visual acuity by manifest refraction of +0.10 logMAR (20/25 Snellen equivalent) or better in each eye.

Exclusion Criteria:

* Regular use of ocular medications (prescription or over-the-counter).
* Current use of systemic medications which, in the investigators opinion, may significantly affect contact lens wear, tear film production, pupil size, accommodation or refractive state.
* Pregnant or lactating or planning a pregnancy at the time of enrolment.
* Known ocular or systemic disease such as, but not limited to: anterior uveitis or iritis, episcleritis or scleritis, glaucoma, Sjogren's syndrome, lupus erythematosus, scleroderma, or diabetes.
* Any ocular, systemic or neuro-developmental conditions that in the investigators opinion, could influence refractive development.
* Keratoconus or an irregular cornea.
* Biomicroscope findings that would contraindicate contact lens wear including, but not limited to:

  1. Any active anterior segment ocular disease that would contraindicate contact lens wear.
  2. clinically significant (Grade 3 or 4) abnormalities of the anterior segment, lids, conjunctiva, sclera or associated structures.
* The investigator for any reason considers that it is not in the best interest of the subject to participate in the study.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, Study Director — Visioncare Research Ltd.
Locations (4):
- University of Waterloo School of Optometry, Waterloo, Ontario, Canada
- University of Minho Clinical & Experiment Optometry Research Lab, Braga, Portugal
- National University of Singapore Faculty of Medicine, Singapore, Singapore
- Aston University Ophthalmic Research Group, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-three participants were enrolled, and 76 participants completed the study. The primary reason was due to decreased vision related to astigmatism.
Units Other Than Participants: Eyes
Groups:
- Dual Focus for 3 Years: Group of subjects who completed dual focus soft contact lens wear treatment for 3 years. Subjects refit to Single Vision Soft Contact Lens for 1 year.
- Dual Focus for 6 Years: Group of subjects who completed dual focus soft contact lens wear treatment for 6 years. Subjects refit to Single Vision Soft Contact Lens for 1 year.
Period: Overall Study
Arm/Group | Dual Focus for 3 Years | Dual Focus for 6 Years
Started | 40; 80 Eyes | 43; 86 Eyes
Completed | 39; 78 Eyes | 37; 74 Eyes
Not Completed | 1; 2 Eyes | 6; 12 Eyes
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Population: Eighty-three participants were enrolled, and demographic data include all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dual Focus for 3 Years | Dual Focus for 6 Years | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (1.58) | 16.3 (1.2) | 16.2 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 20 | 21 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Proportion may not sum to 100% as participants selecting more than one race will be counted multiple times.
  Participants
    Caucasian (European) | 27 | 28 | 55
    East Asian | 10 | 13 | 23
    Indian/Pakistani/SriLankan | 5 | 3 | 8
    Middle Eastern | 1 | 0 | 1
    Hispanic - Latino | 0 | 1 | 1
    Mediterranean | 1 | 0 | 1
    Black British | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Spherical Equivalent Refractive Error (SERE)
Description: Change in spherical equivalent refractive error (SERE) relative to baseline (i.e., at end of dual focus soft contact lens wear treatment of either 3 or 6 years). Cycloplegic autorefraction was used to measure refractive error.
Time Frame: 1 year
Population: [Not specified]
Measure: Mean (Standard Deviation); unit: D
Units Other Than Participants: Eyes
Arm/Group | Dual Focus for 3 Years | Dual Focus for 6 Years
Number analyzed (Participants) | 40 | 43
Number analyzed (Eyes) | 80 | 76
D | -0.23 (0.363) | -0.21 (0.397)

2. Primary Outcome: Change in Axial Length (AL)
Description: Change in axial length (AL) relative to baseline (i.e., at end of dual focus soft contact lens wear treatment of either 3 or 6 years). Partial coherence interferometry was used to measure axial length.
Time Frame: 1 year
Population: [Not Specified]
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Dual Focus for 3 Years | Dual Focus for 6 Years
Number analyzed (Participants) | 40 | 43
Number analyzed (Eyes) | 80 | 76
mm | 0.09 (0.090) | 0.10 (0.103)

ADVERSE EVENTS:
Time Frame: The data was collected in time frame of 1 year of study.
Arm/Group | Dual Focus for 3 Years | Dual Focus for 6 Years
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 2/40 | 3/43
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dual Focus for 3 Years (N=40) | Dual Focus for 6 Years (N=43)
Conjuctivitis (Infections and infestations) | 1 | 1
Corneal Staining (Product Issues) | 1 | 1
Discomfort (Product Issues) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT05779072/Prot_SAP_000.pdf